CLINICAL TRIAL: NCT04253457
Title: The Soft Tissue Injection of Corticosteroid And Local Anaesthetic Study - A Single Site, Non-inferiority Randomised Control Trial Evaluating Pain After Soft Tissue Corticosteroid Injections With and Without Local Anaesthetic
Brief Title: The SToICAL Study - The Soft Tissue Injection of Corticosteroid And Local Anaesthetic Study
Acronym: SToICAL
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Standard of Care change impacted recruitment
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 259336
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Carpal Tunnel Syndrome; De Quervains Tenosynovitis; Trigger Finger
Keywords: Pain VAS Score; Corticosteroid injection; Local anaesthetic
MeSH Terms: conditions — Carpal Tunnel Syndrome; De Quervain Disease; Trigger Finger Disorder | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid injection (Experimental): Single injection of 1ml of triamcinolone (40mg/1ml)
  Interventions: Drug: 1ml of triamcinolone (40mg/1ml)
- Corticosteroid and local anaesthetic injection (Active Comparator): Single injection of 1ml of triamcinolone (40mg/1ml) + 1ml 1% Lidocaine
  Interventions: Drug: 1ml of triamcinolone (40mg/1ml)

INTERVENTIONS:
Drug: 1ml of triamcinolone (40mg/1ml) — Single injection of 1ml of triamcinolone (40mg/1ml)

SUMMARY:
Some hand conditions can be treated with a steroid injection. Some doctors mix the steroid with local anaesthetic in the hope that the patient will experience less pain after the injection. Some doctors do not do this. It is not known if adding local anaesthetic to the steroid improves patient's pain after the injection.

The overall aim of the study is to see whether using local anaesthetic in the steroid injection makes a difference to patients' pain. If the study shows that using local anaesthetic improves patients' pain then the investigators should continue using it. If not, the investigators should stop giving patients unnecessary medication, which would also save the NHS time and money.

DETAILED DESCRIPTION:
This study is a single site, patient and assessor blinded, non-inferiority randomised control trial of patients with a clinical diagnosis of trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome, treated with a corticosteroid injection co-administered with or without local anaesthetic.

The aim is to determine whether pain experienced during the 24 hours after a corticosteroid injection to the hand and wrist is no worse than (not inferior to) the pain experienced after a corticosteroid and local anaesthetic injection.

The primary outcome is to investigate whether there is a difference in pain VAS scores at 1-hour after a corticosteroid injection for trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome co-administered with or without local anaesthetic. Secondary outcomes look at differences in pain VAS scores within the first 24-hours after the injection, at the time of the injection and enquires about effects on hand function.

Patients attending elective hand and wrist outpatient clinics at the University Hospitals Plymouth NHS Trust with a clinical diagnosis of trigger finger, de Quervains tenosynovitis and carpal tunnel syndrome will be screen for eligibility for recruitment.

All patients over the age 18 years old with a clinical diagnosis of trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome and who are able to give written informed consent for treatment will be included. Patients will be excluded if they have had previous surgery or corticosteroid injection for the condition being treated at the site considered for injection. A previous corticosteroid injection elsewhere in the hand does not exclude a patient from the trial. Those who are pregnant, breast-feeding or who have a history of hypersensitivity to corticosteroid or local anaesthetic will be excluded.

The study will run for a 12-month period or until 100 patients have been recruited to the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages >/= 18 years
* A clinical diagnosis of trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome made by a consultant physician.
* Treatment with corticosteroid injection is recommended by the doctor and agreed by the patient
* Patient is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Previous surgery for the condition being treated at the desired location of injection
* Previous steroid injection for the condition being treated at the desired location of injection
* Clinical suspicion of local or systematic sepsis or infection
* History of hypersensitivity to the corticosteroid or local anaesthetic
* Pregnant or breast-feeding females
* Unable to understand and complete self-report questionnaires written in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Pain visual analog scale scores at 1 hour | 1 hour
  Investigate whether there is a difference in pain visual analog scale scores (where 0 is no pain and 10 is the worst pain possible) at 1-hour after a corticosteroid injection for trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome co-administered with or without local anaesthetic.

SECONDARY OUTCOMES:
Pain visual analog scale scores during 24 hours | 24 hours
  Investigate whether there is a difference in pain visual analog scale scores (where 0 is no pain and 10 is the worst pain possible) during the 24-hours after a corticosteroid injection for trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome co-administered with or without local anaesthetic.
Pain visual analog scale score at the time of injection | Immediate
  Investigate whether there is a difference in the pain visual analog scale scores (where 0 is no pain and 10 is the worst pain possible) at the time of the corticosteroid injection for trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome co-administered with or without local anaesthetic.
Pain and functional loss | 3 hours
  Investigate the difference in the additional analgesia required and in the functional use of the hand during the first 3 hours following a corticosteroid injection for trigger finger, de Quervains tenosynovitis or carpal tunnel syndrome co-administered with or without local anaesthetic.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Gozzard, MD, Principal Investigator — University Hospitals Plymouth NHS Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones M, Evans J, Fullilove S, Doyle E, Gozzard C. The SToICAL trial: study protocol for the soft tissue injection of corticosteroid and local anaesthetic trial-a single site, non-inferiority randomised control trial evaluating pain after soft tissue corticosteroid injections with and without local anaesthetic. Trials. 2021 Sep 28;22(1):662. doi: 10.1186/s13063-021-05627-5. PMID 34583762

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04253457/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04253457/ICF_001.pdf